CLINICAL TRIAL: NCT01861418
Title: Effects of Lumbopelvic Manipulation on Neuromuscular Activity of Back and Hip Muscles in Adults With Chronic Low Back Pain
Brief Title: Effects of Lumbopelvic Manipulation on Neuromuscular Activity of Back & Hip Muscles in Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TexasWU
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2016-10

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; low back pain; lumbopelvic manipulation; Chicago manipulation; EMG median frequency; electromyography; reliability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham manipulation (Placebo Comparator): Each participant will lie in a supine position. The treating investigator (TI) will stand on the opposite side of the low back pain. Then, the participant will be asked to clasp his/her hand behind the neck. The TI will side bend the participant's spine towards the non-painful side, reach through the participant's hands and perform a spinal rotation away from the painful side. The TIs other hand will be placed over the anterior superior iliac spine (ASIS) of the painful side. Lastly, the TI will take up the slack and maintain the pressure on the ASIS for 5-10 seconds and ask the participant whether he/she can tolerate the pressure. If the participant can tolerate the pressure for at least 5 seconds. Then, the subjects will be re-positioned to the starting position.
  Interventions: Other: Sham manipulation
- Lumbopelvic Manipulation, Chicago (Experimental): Each participant will lie in supine position. The treating investigator (TI) will stand opposite of the low back pain. Participant will clasp his/her hand behind the neck. TI will side bend the participant's spine toward non-painful side, reach through participant's hands and perform a spinal rotation away from the painful side. TI's other hand will be placed over the anterior superior iliac spine (ASIS) of the painful side. The TI will take up the slack and maintain pressure on the ASIS for 5-10 seconds and ask participant whether he/she can tolerate the pressure. If participant can tolerate the pressure for at least 5 seconds, verbal permission will be obtained from the participant and the TI will proceed and apply a high-velocity low-amplitude posterior thrust force over the ASIS.
  Interventions: Other: Lumbopelvic Manipulation

INTERVENTIONS:
Other: Lumbopelvic Manipulation — Participant will lie in supine position. The treating investigator (TI) will stand on opposite side of low back pain. Participant will clasp his/her hand behind the neck. TI will side bend participant's spine towards non-painful side. TI will reach through participant's hands and perform spinal rotation away from painful side. TI's other hand will be placed over anterior superior iliac spine (ASIS) of painful side. TI will take up the slack and maintain pressure on the ASIS for 5-10 seconds and ask the participant whether he/she can tolerate the pressure. If participant can tolerate the pressure for at least 5 seconds, verbal permission will be obtained from participant and TI will proceed and apply a high-velocity low-amplitude posterior thrust force over the ASIS.
  Other Names: Chicago Manipulation Technique
  Arms: Lumbopelvic Manipulation, Chicago
Other: Sham manipulation — Each participant will be asked to lie in a supine position. The treating investigator will stand on the opposite side of the low back pain. Then, the participant will be asked to clasp his/her hand behind the neck. The treating investigator will side bend the participant's spine towards the non-painful side to mid-range. The treating investigator will reach through the participant's hands and perform a spinal rotation away from the painful side to the mid-range. The treating investigator's other hand will be placed over the anterior superior iliac spine (ASIS) of the painful side.
  Arms: Sham manipulation

SUMMARY:
The purposes of this study are:

1. To examine the within-day and between-day test-retest reliability of a testing protocol measuring the back and hip muscles fatigability using EMG median frequency
2. To examine the immediate and the carry-over effects of the lumbopelvic manipulation on the EMG median frequency of the lumbar multifidus (MULT), gluteus medius (GMED) and gluteus maximus (GMAX) muscles in patients with chronic low back pain (CLBP)
3. To compare the fatigability levels of the MULT, GMED and GMAX muscles by measuring the EMG median frequency between the participants who will receive lumbopelvic manipulation.

The research hypotheses are:

1. The testing protocol using EMG median frequency as a fatigue indicator for MULT,GMED and GMAX muscles will have good (ICC ≥ 0.80) within-day and between-day test-retest reliability.
2. The fatigability level of the MULT, GMED and GMAX muscles will significantly decrease immediately after the lumbopelvic manipulation and will be maintained over two to four days following the manipulation.
3. The fatigability of the MULT, GMED and GMAX muscles will significantly decrease after the intervention in the manipulation group while no change will occur in the placebo group.

ELIGIBILITY:
Healthy subjects or the reliability phase:

Inclusion Criteria:

* Subjects without any history of back problems
* Subjects without any known pathology.

Exclusion Criteria:

* Any serious spinal condition such as tumor, fracture, or infection,
* Signs of nerve root compression (i.e. straight leg- raise ≤ 45° or diminished reflexes, sensation or lower extremity strength),
* Structural deformity,
* Spondylolithesis ,
* Ankylosing spondylitis
* Spinal stenosis,
* Osteoporosis,
* Previous surgery to the back or the hip, and
* Current pregnancy.

Subjects with Chronic low back pain for both the reliability and the manipulation phases:

Inclusion Criteria:

* Participants should be between the age of 20 to 60 years.
* Have had complaints of chronic low back pain for at least three months.

Exclusion Criteria:

* Any serious spinal condition such as tumor, fracture, or infection,
* Signs of nerve root compression (i.e. straight leg- raise ≤ 45° or diminished reflexes, sensation or lower extremity strength),
* Structural deformity,
* Spondylolithesis ,
* Ankylosing spondylitis
* Spinal stenosis,
* Osteoporosis,
* Previous surgery to the back or the hip, and
* Current pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Amount of Change in Muscles Endurance | Baseline, Immediately, 15-minutes, 30-minutes, and two to four days after the intervention
  electromyographic (EMG) median frequency will be used to determine the endurance of the gluteus maximums, gluteus medius and the lumbar multifidus muscles. The EMG median frequency will be measured in Hertz (Hz).

SECONDARY OUTCOMES:
Amount of Change in Pain Level | Baseline, immediately, 15-minutes, 30-minutes, and two to four days after the intervention
  Pain Visual Analogue Scale (VAS) will be used in this study. Participants will be asked to rate their pain level on a 10-cm horizontal line which is marked on the left end "No pain" and on the right end "Extreme pain". Then, the pain level for a specific participant will be determined by measuring the line from the "No pain" end to the mark placed by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A Almadan, PhD Student, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States